CLINICAL TRIAL: NCT05082571
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of Once Daily Oral Vadadustat for the Treatment of Pediatric Subjects With Anemia of Chronic Kidney Disease After Conversion From an Erythropoiesis-stimulating Agent
Brief Title: Study to Evaluate the Safety and Efficacy of Oral Vadadustat in Pediatric Participants With Anemia of Chronic Kidney Disease
Acronym: CONVERSION
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0041
Record Dates: First submitted 2021-09-28; First posted 2021-10-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: anemia; kidney disease; vadadustat; pediatric population; children; chronic kidney disease; erythropoiesis stimulating agent; dialysis; hypoxia-inducible factor (HIF) prolyl hydroxylase inhibitor
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic | interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vadadustat (Experimental): Cohort 1: participants with ≥12 years to <17 years; Cohort 2: participants with ≥6 years to <12 years; Cohort 3(a): participants with ≥2 years to <6 years; and Cohort 3(b): participants with ≥4 months to <2 years
  Interventions: Drug: vadadustat

INTERVENTIONS:
Drug: vadadustat — Vadadustat tablet orally once a day for 52 weeks
  Other Names: AKB-6548

SUMMARY:
This study will assess the safety and efficacy of once daily dosing of vadadustat for the treatment of pediatric participants with anemia of Chronic Kidney Disease (CKD) after conversion from an Erythropoiesis Stimulating Agent (ESA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anemia of chronic kidney disease (CKD)
* Diagnosis of non-dialysis-dependent (NDD) CKD with an estimated glomerular filtration rate of greater than (>) 10 and less than (<) 60 milliliters/minute/1.73 meters^2 (mL/min/1.73 m^2) or diagnosis of dialysis dependent (DD) CKD
* Mean hemoglobin (Hb) between 9.0 and 12.0 grams/deciliters (g/dL) (inclusive)
* Transferrin Saturation ≥ 20%

Exclusion Criteria:

* Anemia due to a cause other than CKD
* Active bleeding or recent clinically significant blood loss
* History of sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red Blood Cells transfusion within 4 weeks
* Serum albumin level less than 2.5 g/dL
* Uncontrolled hypertension
* Active malignancy or treatment for malignancy within the past 2 years prior to Screening
* Evidence of iron overload or diagnosis of hemochromatosis
* Known hypersensitivity to vadadustat or any excipients in vadadustat tablet

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Hemoglobin (Hb) Values Between Baseline and the Primary Evaluation Period (Average Hb From Weeks 21 to 28) | Baseline; Weeks 21 to 28

SECONDARY OUTCOMES:
Time to Achieve Hb Levels of ≥10.0 grams/deciliters (g/dL) | Up to Week 52
Number of Participants With Mean Hb Values Within the Target Range During the Primary Evaluation Period | From Week 21 to Week 28
Number of Participants With Mean Hb Values Within the Target Range During the Extension Period | From Week 29 to Week 52
Number of Participants With Treatment-emergent Adverse Events and who Discontinued From the Study due to Adverse Events | Up to Week 56
Maximum Observed Plasma Concentration (Cmax) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Time to Reach Cmax (Tmax) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC 0-t) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Terminal Elimination Half-Life (t1/2) of Vadadustat and its Metabolites | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Serum Erythropoietin (EPO) | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Reticulocyte Count | Pre-dose and post-dose at intermediate time points up to 28 weeks
Change From Baseline in Hb levels | Pre-dose and post-dose at intermediate time points up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (1):
- Research Site, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No